CLINICAL TRIAL: NCT01633112
Title: A 12-month, Randomized, Rater- and Dose-blinded Study to Compare the Efficacy and Safety of Fingolimod 0.25 mg and 0.5 mg Administered Orally Once Daily With Glatiramer Acetate 20 mg Administered Subcutaneously Once Daily in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: MS Study Evaluating Safety and Efficacy of Two Doses of Fingolimod Versus Copaxone
Acronym: ASSESS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720D2312
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-04

CONDITIONS: Relapsing-remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride; Glatiramer Acetate; Coat Protein Complex I

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Fingolimod patients were dose blind.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fingolimod 0.5 mg (Experimental): orally once daily
  Interventions: Drug: fingolimod
- fingolimod 0.25mg (Experimental): orally once daily
  Interventions: Drug: fingolimod
- glatiramer acetate 20 mg (Active Comparator): subcutaneous once daily
  Interventions: Drug: glatiramer acetate

INTERVENTIONS:
Drug: fingolimod — capsule
  Other Names: FTY720, fingolimod hydrochloride,; Gilenya
  Arms: fingolimod 0.25mg; fingolimod 0.5 mg
Drug: glatiramer acetate — subcutaneous injection
  Other Names: Copaxone, Glatopa
  Arms: glatiramer acetate 20 mg

SUMMARY:
The purpose of this study was to demonstrate that at least one dose (0.5 mg followed by 0.25 mg) of fingolimod is superior to glatiramer acetate 20 mg SC in reducing the ARR up to 12 months in patients with relapsing-remitting MS

DETAILED DESCRIPTION:
This was a multicenter, randomized, rater- and dose-blinded, study to compare the efficacy and safety of 0.25 mg and 0.5 mg of fingolimod with glatimer acetate 20 mg s.c. in patients with RRMS.

This study consisted of 3 periods:

* Screening Period: up to 45 days for all patients
* Treatment Period: 12 months of glatiramer acetate 20 mg, fingolimod 0.25 mg, or fingolimod 0.5 mg
* Follow-up occurred 3 months (12 weeks) after the last dose of study drug for all patients The informed consent form was signed prior to any study related activities at the screening visit. Randomization to either treatment group was preformed at visit 1 after a diligent check of applicable in- and exclusion criteria in a 1:1:1 ratio (changed to 5:3:2 after implementation of Amendment 2 in 2015).

Treatment groups:

* fingolimod 0.5 mg/day orally for up to 12 months
* fingolimod 0.25 mg/day orally for up to 12 months
* glatiramer acetate 20 mg/day subcutaneously for up to 12 months

ELIGIBILITY:
Inclusion criteria:

* Written informed consent must be obtained before any assessment is performed
* Male and female patients 18 to 65 years of age, inclusive.
* Patients with RRMS, as defined by 2010 revised McDonald criteria.
* Patients must be neurologically stable with no onset of relapse within 30 days of randomization
* Patients with at least 1 documented relapse during the previous year or 2 documented relapses during the previous 2 years before randomization.
* Patients with an EDSS score of 0 to 6, inclusive, at Screening. A score of 6.0 indicates unilateral assistance (cane or crutch) required to walk at least 100 meters with or without resting.

Exclusion criteria:

* Patients with a history of malignancy of any organ system (other than cutaneous basal cell carcinoma) in the last 5 years that do not have confirmation of absence of a malignancy prior to randomization
* Patients with an active chronic disease (or stable but treated with immune therapy) of the immune system other than MS (e.g., rheumatoid arthritis, scleroderma, Sjogren's syndrome, Crohn's disease, ulcerative colitis) or with a known immunodeficiency syndrome (HIV-antibody positive, AIDS, hereditary immune deficiency, drug-induced immune deficiency).
* Patients who have been treated with:
* High-dose intravenous (IV) immunoglobulin (Ig) within 4 weeks before randomization
* Immunosuppressive/chemotherapeutic medications (e.g., azathioprine, cyclophosphamide, methotrexate) within 6 months before randomization
* Natalizumab within 2 months before randomization
* Previous treatment with lymphocyte-depleting therapies (e.g., rituximab, alemtuzumab, ofatumumab, ocrelizumab, or cladribine) within 1 year before randomization Previous treatment with mitoxantrone within 6 months before randomization
* Use of teriflunomide within 3.5 months prior to randomization, except if active washout (with either cholestyramine or activated charcoal) was done. In that case, plasma levels are required to be measured and be below 0.02 mg/L before randomization.

No washout period is necessary for patients treated with dimethyl fumarate, interferon (IFN) beta, or glatiramer acetate.

Patients being treated with dimethyl fumarate, glatiramer acetate, or IFN beta at the Screening visit can continue drug intake up to the day before Day 1 of this study (i.e., there is no need for a washout period).

* Patients who have been treated with systemic corticosteroids or adrenocorticotropic hormones in the past 30 days prior to the screening magnetic resonance imaging (MRI) procedure.
* Patients with uncontrolled diabetes mellitus (glycosylated hemoglobin >9%) or with diabetic neuropathy.
* Patients with a diagnosis of macular edema during Screening (patients with a history of macular edema will be allowed to enter the study provided that they do not have macular edema at Screening).
* Patients with severe active bacterial, viral, or fungal infections.
* Patients without acceptable evidence of immunity to varicella zoster virus (VZV) at randomization.
* Patients who have received any live or live-attenuated vaccines (including VZV, herpes simplex, or measles) within 1 month before randomization.
* Patients who have received total lymphoid irradiation or bone marrow transplantation.
* Patients with any unstable medical/psychiatric condition, as assessed by the primary treating physician at each site.
* Patients who in the last 6 months experienced any of the following cardiovascular conditions or findings in the screening electrocardiogram (ECG): myocardial infarction, unstable angina, stroke, transient ischemic attack or decompensated heart failure requiring hospitalization or Class III/IV heart failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1064 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (117):
- United States (91):
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Loveland, Colorado
  - Novartis Investigative Site, Fairfield, Connecticut
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Naples, Florida
  - Novartis Investigative Site, New Port Richey, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Pompano Beach, Florida
  - Novartis Investigative Site, Ponte Vedra Beach, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Elk Grove Village, Illinois
  - Novartis Investigative Site, Evanston, Illinois
  - Novartis Investigative Site, Flossmoor, Illinois
  - Novartis Investigative Site, Northbrook, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, West Des Moines, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Hammond, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Farmington Hills, Michigan
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Traverse City, Michigan
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Teaneck, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Amherst, New York
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Patchogue, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Stony Brook, New York
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Bellevue, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Cordova, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Round Rock, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sherman, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Alexandria, Virginia
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Roanoke, Virginia
  - Novartis Investigative Site, Issaquah, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Brazil (9):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Campina Grande do Sul
  - Novartis Investigative Site, Goiânia
  - Novartis Investigative Site, Passo Fundo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Canada (6):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Santiago, Chile
- Mexico (7):
  - Novartis Investigative Site, Tlalnepantla, Edo de Mexico
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Chihuahua City
  - Novartis Investigative Site, Monterrey
- Novartis Investigative Site, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Cree BAC, Goldman MD, Corboy JR, Singer BA, Fox EJ, Arnold DL, Ford C, Weinstock-Guttman B, Bar-Or A, Mientus S, Sienkiewicz D, Zhang Y, Karan R, Tenenbaum N; ASSESS Trial Investigators. Efficacy and Safety of 2 Fingolimod Doses vs Glatiramer Acetate for the Treatment of Patients With Relapsing-Remitting Multiple Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2020 Aug 24;78(1):1-13. doi: 10.1001/jamaneurol.2020.2950. Online ahead of print. PMID 32852530

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1461 subjects were screened for participation in this study; of those, 1064 subjects were randomly assigned to study treatment
Groups:
- FTY720 0.5 mg: Fingolimod (FTY720) 0.5 mg orally once a day for up to 12 months
- FTY720 0.25 mg: Fingolimod (FTY720) 0.25 mg orally once a day for up to 12 months
- GA 20 mg: Glatiramer acetate (GA) 20 mg s.c. once a day for up to 12 months
Period: Overall Study
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Started | 352 | 370 | 342
Completed | 299 | 310 | 250
Not Completed | 53 | 60 | 92
Not completed — Lack of Efficacy | 1 | 6 | 13
Not completed — Abnormal laboratory value(s) | 3 | 1 | 0
Not completed — Abnormal test procedure result(s) | 0 | 1 | 0
Not completed — Administrative problems | 1 | 2 | 5
Not completed — Adverse Event | 16 | 18 | 20
Not completed — Lost to Follow-up | 7 | 19 | 6
Not completed — Protocol Violation | 4 | 0 | 2
Not completed — Subject no longer requires study drug | 0 | 0 | 1
Not completed — Withdrawal by Subject | 20 | 12 | 41
Not completed — missing Study Completion CRF | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Ramdomized set: All subjects who were assigned randomization numbers. The subjects in this set were called randomized subjects. This set was used to summarize subject disposition, demographic and baseline characteristics, and protocol deviation information. Subjects were grouped according to randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg | Total
Number analyzed (Participants) | 352 | 370 | 342 | 1064
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (11.12) | 38.9 (11.01) | 39.6 (10.80) | 39.6 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264 | 276 | 252 | 792
  Male | 88 | 94 | 90 | 272
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 268 | 279 | 243 | 790
  Black | 34 | 43 | 41 | 118
  Asian | 0 | 1 | 0 | 1
  Native American | 8 | 7 | 9 | 24
  Pacific Islander | 0 | 1 | 0 | 1
  Other | 42 | 39 | 49 | 130

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Annualized Relapse Rate
Description: Annualized relapse rate (ARR) was defined as the average number of confirmed relapses per year (i.e., the total number of confirmed relapses divided by the total days in the study multiplied by 365.25). The number of relapses included all the confirmed relapses experienced during the study from first dose to end of study.
Time Frame: up to 12 months
Population: Full-analysis set: All subjects who were randomly assigned and took at least 1 dose of study drug. Following the intent-to-treat principle, subjects were grouped according to the assigned treatment at randomization. Efficacy analyses were performed using the full analysis set unless otherwise notified.
Measure: Number (95% Confidence Interval); unit: relapses/year
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
relapses/year | 0.153 [0.111 to 0.212] | 0.221 [0.168 to 0.290] | 0.258 [0.196 to 0.341]
Statistical Analysis 1: Comparison: FTY720 0.5 mg vs GA 20 mg; H01: µ FTY 0.5 mg = µ GA versus HA1: µ FTY 0.5 mg ≠µ GA H02: µ FTY 0.25 mg = µ GA versus HA2: µ FTY 0.25 mg ≠µ GA; Test type: Superiority — For each of the 2 FTY720 doses, the null hypothesis was that there was no difference in the ARRs between subjects treated with FTY720 and those treated with GA versus the alternative hypothesis that there was a difference between the 2 treatment arms. In order to preserve the Type I experiment-wise error rate, the null hypothesis was rejected if the observed p-value for the between-treatment comparison was less than the significance level as specified in the multiplicity adjustment procedure; p = 0.0138, negative binomial regression model; adjusted for treatment, geographical region, number of relapses in the previous year, baseline EDSS, and baseline Gd-enhancing T1 lesion count
Statistical Analysis 2: Comparison: FTY720 0.25 mg vs GA 20 mg; H01: µ FTY 0.5 mg = µ GA versus HA1: µ FTY 0.5 mg ≠µ GA H02: µ FTY 0.25 mg = µ GA versus HA2: µ FTY 0.25 mg ≠µ GA; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4153, negative binomial regression model; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: New or Newly Enlarging T2 Lesions
Description: Inflammatory activity based on MRI measurement of new/newly enlarged T2 lesion count.
Time Frame: At 12 months/end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
Lesions | 2.6 (5.42) | 3.3 (6.94) | 5.7 (10.71)
Statistical Analysis 1: Comparison: FTY720 0.5 mg vs GA 20 mg; Test type: Other; p < 0.0001, negative binomial regression model; Adjusted for treatment, geog. region, age, baseline T2 lesion count, baseline Gd-enhancing T1 lesion count, and the number of previous year relapses
Statistical Analysis 2: Comparison: FTY720 0.25 mg vs GA 20 mg; Test type: Other; p < 0.0001, negative binomial regression model; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Participants Free of New/Newly Enlarged T2 Lesions
Description: Inflammatory activity based on MRI measurement of new/newly enlarged T2 lesion count.
Time Frame: At 12 months/end of study
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
Participants | 156 | 155 | 96

4. Secondary Outcome: Change From Baseline in T2 Lesion Volume
Description: Inflammatory activity based on MRI measurement of new/newly enlarged T2 lesion volume
Time Frame: Baseline, 12 months/end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic centimeters (cc)
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
cubic centimeters (cc) | -0.14 (1.583) | -0.05 (2.340) | 0.42 (2.305)
Statistical Analysis 1: Comparison: FTY720 0.5 mg vs GA 20 mg; Test type: Other; p < 0.0001, ANCOVA; rank ANCOVA with covariates: adjusted for treatment, age, region, number of relapses experienced in the previous year, and baseline T2 lesion volume
Statistical Analysis 2: Comparison: FTY720 0.25 mg vs GA 20 mg; Test type: Other; p = 0.0060, ANCOVA; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Gd Enhancing T1 Lesion Count
Description: Inflammatory activity based on MRI measurement of Gd enhancing T1 lesion count
Time Frame: At 12 months/end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
lesions | 0.4 (1.57) | 0.4 (1.56) | 0.9 (3.67)
Statistical Analysis 1: Comparison: FTY720 0.5 mg vs GA 20 mg; Test type: Other; p = 0.0167, negative binomial regression model; adjusted for treatment, age, geog. region, baseline T2 lesion count, baseline Gd-enhancing T1 lesion count, and the number of previous year relapses
Statistical Analysis 2: Comparison: FTY720 0.25 mg vs GA 20 mg; Test type: Other; p = 0.0011, negative binomial regression model; adjusted for treatment, age, geog. region, baseline T2 lesion count, baseline Gd-enhancing T1 lesion count, and the number of previous year relapses

6. Secondary Outcome: Gd Enhancing T1 Lesion Volume
Description: Inflammatory activity based on MRI measurement of Gd enhancing T1 lesion count
Time Frame: Baseline, 12 months/end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic centimeter
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
cubic centimeter
  Baseline: number analyzed (Participants) | 343 | 364 | 322
  Baseline | 0.31 (1.067) | 0.32 (1.421) | 0.22 (0.841)
  Month 12/end of study: number analyzed (Participants) | 302 | 325 | 263
  Month 12/end of study | 0.06 (0.215) | 0.05 (0.181) | 0.12 (0.450)
Statistical Analysis 1: Comparison: FTY720 0.5 mg vs GA 20 mg; Test type: Other; p = 0.0052, ANCOVA; ranked ANCOVA with covariates: treatment, region, age, baseline Gd-enhancing T1 lesion volume, and number ofrelapses experienced in the previous year
Statistical Analysis 2: Comparison: FTY720 0.25 mg vs GA 20 mg; Test type: Other; p = 0.0636, ANCOVA; [statistical method as in outcome 6, analysis 1]

7. Secondary Outcome: Percentage of Patients Free of New T1 Hypointense Lesions
Description: Based on MRI measures of new T1 hypointense lesions
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
Percentage | 55.3 | 52.1 | 44.3
Statistical Analysis 1: Comparison: FTY720 0.5 mg vs GA 20 mg; Test type: Other; p = 0.0011, Regression, Logistic — adjusted for treatment, region, age, proper baseline T1 lesion variable, baseline Gd-enhancing T1 lesion count and number of previous year relapses; pair-wise comparisons between treatment groups using a logistic regression model
Statistical Analysis 2: Comparison: FTY720 0.25 mg vs GA 20 mg; Test type: Other; p = 0.0146, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; pair-wise comparisons between treatment groups using a logistic regression model

8. Secondary Outcome: Change From Baseline in TSQM Scales
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) was developed and validated as a general measure for treatment satisfaction. Each scale score was calculated by summing individual items and then transformed to a 0-100 scale. Higher summary scores indicate better satisfaction with study drug.
Time Frame: 6 months, 12 months/end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
score on a scale
  Global Satisfaction (Month 6): number analyzed (Participants) | 175 | 200 | 153
  Global Satisfaction (Month 6) | 20.8 (28.15) | 23.4 (27.04) | 14.4 (25.42)
  Global Satisfaction (Month 12): number analyzed (Participants) | 185 | 201 | 180
  Global Satisfaction (Month 12) | 19.2 (31.87) | 20.5 (32.21) | 9.4 (30.43)
  Effectiveness (Month 6): number analyzed (Participants) | 176 | 197 | 151
  Effectiveness (Month 6) | 15.2 (25.96) | 18.2 (25.05) | 12.9 (23.43)
  Effectiveness (Month 12): number analyzed (Participants) | 187 | 198 | 178
  Effectiveness (Month 12) | 16.8 (26.85) | 17.9 (28.29) | 8.0 (27.38)
  Side Effects (Month 6): number analyzed (Participants) | 173 | 196 | 149
  Side Effects (Month 6) | 16.9 (31.58) | 18.8 (30.63) | 9.3 (31.94)
  Side Effects (Month 12): number analyzed (Participants) | 185 | 194 | 174
  Side Effects (Month 12) | 16.2 (31.52) | 17.2 (32.52) | 7.6 (32.76)
  Convenience (Month 6): number analyzed (Participants) | 176 | 197 | 151
  Convenience (Month 6) | 30.7 (25.76) | 26.5 (25.93) | 4.4 (20.73)
  Convenience (Month 12): number analyzed (Participants) | 187 | 198 | 178
  Convenience (Month 12) | 29.5 (24.42) | 26.5 (26.36) | 0.8 (25.72)
Statistical Analysis 1: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Global Satisfaction (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 2: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Global Satisfaction (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 3: Comparison: GA 20 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Global Satisfaction (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 4: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Global Satisfaction (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 5: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Global Satisfaction (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 6: Comparison: GA 20 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Global Satisfaction (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 7: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Effectiveness (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 8: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Effectiveness (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 9: Comparison: GA 20 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Effectiveness (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 10: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Effectiveness (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 11: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Effectiveness (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 12: Comparison: GA 20 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Effectiveness (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 13: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Side Effects (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 14: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Side Effects (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 15: Comparison: GA 20 mg; Test type: Other; p = 0.0005, Wilcoxon signed-rank test; Side Effects (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 16: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0051, Wilcoxon signed-rank test; Side Effects (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 17: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Side Effects (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 18: Comparison: GA 20 mg; Test type: Other; p = 0.0051, Wilcoxon signed-rank test; Side Effects (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 19: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Convenience (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 20: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Convenience (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 21: Comparison: GA 20 mg; Test type: Other; p = 0.0068, Wilcoxon signed-rank test; Convenience (Month 6): p-values for within treatment comparison from baseline
Statistical Analysis 22: Comparison: FTY720 0.5 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Convenience (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 23: Comparison: FTY720 0.25 mg; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Convenience (Month 12): p-values for within treatment comparison from baseline
Statistical Analysis 24: Comparison: GA 20 mg; Test type: Other; p = 0.4595, Wilcoxon signed-rank test; Convenience (Month 12): p-values for within treatment comparison from baseline

9. Secondary Outcome: Percent Brain Volume Change From Baseline
Description: Using a Central MRI vendor to ensure calibrated MRI scanning equipment across all sites, MRI scans were performed on subjects following the established parameters and transferred to the central vendor for review of quality and assessment/evaluation.
Time Frame: Baseline, 12 months, end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentages of volume change
Arm/Group | FTY720 0.5 mg | FTY720 0.25 mg | GA 20 mg
Number analyzed (Participants) | 345 | 366 | 324
Percentages of volume change | -0.652 (0.7810) | -0.636 (0.8097) | -0.561 (0.7819)
Statistical Analysis 1: Comparison: FTY720 0.5 mg vs GA 20 mg; Test type: Other; p = 0.1045, ANCOVA; rank ANCOVA model adjusted for treatment, region, age, the number of relapses experienced in the previous year, and baseline normalized brain volume
Statistical Analysis 2: Comparison: FTY720 0.25 mg vs GA 20 mg; Test type: Other; p = 0.1358, ANCOVA; [statistical method as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious AEs (SAEs) were collected during treatment exposure and follow up where: AE summaries on the follow-up set were conducted for time periods defined by days relative to study drug discontinuation: days 1 - 45 after discontinuation, or day 46 or later after drug discontinuation. For SAEs (death and non-fatal ), all SAEs starting after the first dose date, including those starting > 45 days after study drug discontinuation, were included in the safety set summaries.
Groups:
- Fingolimod 0.5 mg: Fingolimod (FTY720) 0.5 mg orally once a day for up to 12 months
- FTY 0.25 mg: Fingolimod (FTY720) 0.25 mg orally once a day for up to 12 months
- All@Patients: All patients in the trial
Arm/Group | Fingolimod 0.5 mg | FTY 0.25 mg | GA 20 mg | All@Patients
All-Cause Mortality (participants affected / at risk) | 0/345 | 0/366 | 0/324 | 0/1035
Serious Adverse Events (participants affected / at risk) | 25/345 | 32/366 | 20/324 | 77/1035
Other Adverse Events (participants affected / at risk) | 214/345 | 245/366 | 190/324 | 649/1035
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=345) | FTY 0.25 mg (N=366) | GA 20 mg (N=324) | All@Patients (N=1035)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Chest pain (General disorders) | 1 | 0 | 0 | 1
Feeling cold (General disorders) | 1 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 2
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1
Extradural abscess (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Meningitis fungal (Infections and infestations) | 0 | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 5
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 0 | 7
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1
Cranial nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 3 | 0 | 4
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 4 | 7 | 7 | 18
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 2 | 0 | 3
Syncope (Nervous system disorders) | 0 | 0 | 2 | 2
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=345) | FTY 0.25 mg (N=366) | GA 20 mg (N=324) | All@Patients (N=1035)
Lymphopenia (Blood and lymphatic system disorders) | 23 | 18 | 1 | 42
Diarrhoea (Gastrointestinal disorders) | 21 | 23 | 10 | 54
Nausea (Gastrointestinal disorders) | 24 | 30 | 15 | 69
Fatigue (General disorders) | 46 | 46 | 22 | 114
Injection site erythema (General disorders) | 0 | 0 | 34 | 34
Injection site pain (General disorders) | 0 | 0 | 36 | 36
Injection site pruritus (General disorders) | 0 | 0 | 26 | 26
Injection site reaction (General disorders) | 0 | 0 | 21 | 21
Nasopharyngitis (Infections and infestations) | 23 | 23 | 14 | 60
Upper respiratory tract infection (Infections and infestations) | 30 | 35 | 20 | 85
Urinary tract infection (Infections and infestations) | 44 | 43 | 35 | 122
Alanine aminotransferase increased (Investigations) | 20 | 15 | 4 | 39
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 20 | 13 | 48
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 19 | 18 | 54
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 24 | 17 | 65
Dizziness (Nervous system disorders) | 12 | 27 | 14 | 53
Headache (Nervous system disorders) | 51 | 50 | 27 | 128
Anxiety (Psychiatric disorders) | 13 | 21 | 9 | 43
Depression (Psychiatric disorders) | 23 | 19 | 18 | 60
Insomnia (Psychiatric disorders) | 12 | 27 | 9 | 48
Hypertension (Vascular disorders) | 26 | 34 | 12 | 72

LIMITATIONS AND CAVEATS:
Terminated due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT01633112/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT01633112/SAP_001.pdf